CLINICAL TRIAL: NCT04268251
Title: Prospective MRI Evaluation of Cavernous Sinus Invasion by Pituitary Adenoma Using Deep Learning Based Denoising
Brief Title: Evaluation of Cavernous Sinus Invasion by Pituitary Adenoma Using Deep Learning Based Denoising MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Sung Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AsanMCHSKim_06
Record Dates: First submitted 2020-01-13; First posted 2020-02-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cavernous Sinus Invasion by Pituitary Adenoma
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep learning based denoising MR (Experimental): 1 mm slice thickness coronal contrast-enhanced T1 weighted imaging with deep learning based denoising vs. 3 mm slice thickness coronal contrast-enhanced T1 weighted imaging
  Interventions: Diagnostic Test: MRI with deep learning based denoising

INTERVENTIONS:
Diagnostic Test: MRI with deep learning based denoising — 1-mm coronal contrast-enhanced T1 weighted image with deep learning based denoising

SUMMARY:
Preoperative evaluation of cavernous sinus invasion by pituitary adenoma is critical for performing safe operation and deciding on surgical extent as well as for treatment success. Because of the small size of the pituitary gland and sellar fossa, determining the exact relationship between the pituitary adenoma and cavernous sinus can be challenging. Performing thin slice thickness MRI may be beneficial but is inevitably associated with increased noise level. By applying deep learning based denoising algorithm, diagnosis of cavernous sinus invasion by pituitary adenoma may be improved.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing preoperative brain MR for pituitary adenoma

Exclusion Criteria:

* Patients who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulates, electronic infusion pumps, etc), because such devices may be displaced or malfunction
* Patients who are pregnant or breast feeding; urine pregnancy test will be performed on women of child bearing potential
* Poor MRI image quality due to artifacts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Cavernous sinus invasion | Within 1 week
  Presence or absence of cavernous sinus invasion determined surgically

SECONDARY OUTCOMES:
Size of pituitary adenoma (in mm), laterality of pituitary adenoma (unilateral or bilateral) on the MRI | Within 1 week
  Size of the tumor (in mm), laterality of the tumor (unilateral or bilateral) on the MRI
Margin of pituitary adenoma (well-delineated, poorly delineated) on the MRI | Within 1 week
  Margin of pituitary adenoma (well-delineated, poorly delineated) on the MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sung Kim, MD PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim M, Kim HS, Park JE, Park SY, Kim YH, Kim SJ, Lee J, Lebel MR. Thin-Slice Pituitary MRI with Deep Learning-Based Reconstruction for Preoperative Prediction of Cavernous Sinus Invasion by Pituitary Adenoma: A Prospective Study. AJNR Am J Neuroradiol. 2022 Feb;43(2):280-285. doi: 10.3174/ajnr.A7387. Epub 2022 Jan 6. PMID 34992127